CLINICAL TRIAL: NCT02831374
Title: Assessment Effectiveness of Platelet Rich Plasma in Wound Healing After Surgical Removal of Mandibular Third Molars: A Clinical Study
Brief Title: Effectiveness of Platelet Rich Plasma in Wound Healing
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Linyi People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Ming Shi, Dr, Linyi People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LinyiPH
Record Dates: First submitted 2016-06-23; First posted 2016-07-13 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Impacted Third Molar Tooth
MeSH Terms: interventions — Anesthesia, Local; Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Use of platelet rich plasma (Group A)' (Experimental): Local anesthesia, surgical extraction of impacted third molar, Preparation of PRP gel, Placing platelet Rich plasma and suturing, Postoperative medication
  Interventions: Drug: Local anesthesia; Procedure: surgical extraction of impacted third molar; Biological: Preparation of PRP gel; Procedure: Placing platelet Rich plasma and suturing; Drug: Postoperative medication
- surgical extraction (Group B) (Placebo Comparator): Local anesthesia, surgical extraction of impacted third molar, Suturing, Postoperative medication
  Interventions: Drug: Local anesthesia; Procedure: surgical extraction of impacted third molar; Procedure: Suturing; Drug: Postoperative medication

INTERVENTIONS:
Drug: Local anesthesia — The surgical extraction under local anesthesia (2% Lignocaine and 1:100000 Adrenaline) procedure was the same in all patients.
Procedure: surgical extraction of impacted third molar — After achieving Local anesthesia using 2% lignocaine hydrochloride with 1:100,000 epinephrine, standard Terrence Ward's incision was placed to raise a full thickness mucoperiosteal flap. Disto-buccal bone was carefully exposed and bone surrounding the buccal aspect of impacted tooth was performed using surgical bur under copious irrigation with 0.9% saline. Tooth was elevated using Coupland elevator and if required situations tooth was sectioned with surgical bur to facilitate its removal. The socket was checked for any tooth or bony debris. The bony margins smoothened using a file and irrigated with 0.9% saline.
Biological: Preparation of PRP gel — Before surgery, 10 milliliter of venous blood was collected from the anticubital fossa of the patients forearm and stored into sterile tubes containing anticoagulant (0.5 milliliter citrate phosphate dextrose) from each patient in the experimental group using routine venipuncture procedure. The whole blood is then centrifuged at 1,200 rotations per minute for ten minutes. The supernatant layer obtained was platelet poor plasma and buffy coat was collected in a new sterile tube and centrifuged again at 1,000 rotations per minute for 10 min. The upper half of the supernatant is removed and the lower half is mixed carefully to get platelet rich plasma. Five drops of mixture of 10 % CaCl2 and 1000 Units bovine thrombin to 2 milliliter Platelet rich plasma to obtain the gel form.
  Arms: Use of platelet rich plasma (Group A)'
Procedure: Placing platelet Rich plasma and suturing — Subsequently, platelet rich plasma gel was placed into the extraction sockets of patients in the group A and wound closure was done using simple interrupted 3.0 black silk sutures.
  Arms: Use of platelet rich plasma (Group A)'
Procedure: Suturing — Wound closure was done using simple interrupted 3.0 black silk sutures.
  Arms: surgical extraction (Group B)
Drug: Postoperative medication — Patients were advised regular post extraction and prescribed 500 milligram of paracetemol postoperatively (1 tablet every 6 hours for 2 days).

SUMMARY:
Purpose: This prospective randomized comparative clinical study was conducted to assess the effect of platelet-rich plasma (PRP) gel on soft tissue healing and bone regeneration potential on lower third molar extraction sockets.

Methods: For the study, 50 Patients (37 male, 13 female) requiring surgical removal of a lower impacted third molar and who fulfilled the inclusion criteria were recruited. The patients were categorized into two groups, Group A and Group B. For each group 25 patients were randomly allocated. The predictor variable in Group A was the application of PRP Gel whereas in Group B had no PRP. Postoperative pain, swelling, trismus, soft tissue healing and osseous regeneration was assessed using standard methods. These outcome variables were assessed on 1, 3-, 5-, 7-, and 14-postoperative day. Patients were recalled at the 4th, 10th, and 16th postoperative week for assessment of bone healing. The data were recorded and tabulated.

DETAILED DESCRIPTION:
The study is designed as a prospective randomized comparative clinical study. The sample population was composed of fifty consecutive patients who needed surgical extraction of lower third molar under local anesthesia. The study included 37 male and 13 female with age ranging from 20 to 40 years. All Patients were categorized into GROUP A (wound in which PRP is placed) and GROUP B (socket without PRP). The patients were allocated randomly to each group equally by single-blind technique, irrespective of age and sex.

Ethical approval was obtained from the Institutional Ethics Committee prior to the beginning of the study. The signed consent form obtained from all the patients after explaining the risks and benefits of the surgical procedure. The group A (test group) received topical application of PRP, whereas the group B (control group) was left to heal without PRP.

Clinical assessment:

Postoperative pain was assessed using a 10-point visual analog scale (VAS) with a score of 0 equals "no pain" and 10 equals "very severe pain" Facial swelling was assessed by modification of Schultze-Mosgau et al method, and this involved measuring the length from the tragus to the oral commissure and tragus to the pogonion. The arithmetic sum of the two measurements was considered as facial swelling at the time point. The maximum distance between the maxillary central incisors and the mandibular central incisors was taken as mouth opening. The difference between postoperative and preoperative mouth opening value was considered as trismus. Assessment of soft tissue healing was based on the criteria given by Landry et al. and Gonshor et al. Third molar sockets were assessed radiographically for bone healing by modification of Kelley's method as described by Olufemi et al. The percentage of facial swelling and mouth opening was estimated using the method described by Ogundipe et al.

Protocol for preparation of PRP gel Under all aseptic conditions, PRP was processed by means of a modification of the method of Sonnleitner et al. Before surgery, 10 mL of venous blood was collected from the antecubital fossa of the patient's forearm and stored into sterile tubes containing anticoagulant (0.5 mL citrate phosphate dextrose) from each patient of group A in the experimental group using routine venipuncture procedure. The tube was thoroughly agitated to ensure mixing of anticoagulant with the venous blood. The whole blood is then centrifuged at 1,200 rpm for ten minutes. The supernatant layer obtained was platelet poor plasma (PPP) and Buffy coat (BC) and RBCs (red blood cells) at the bottom part. PPP, BC and upper 1-2 mm of RBC (red blood cell) layer was collected in a new sterile tube and centrifuged again at 1,000 rpm for 10 min. The upper half of the supernatant is removed and the lower half is mixed carefully to get PRP. The platelet concentration of the PRP was noted.

PRP gel was prepared by adding Five drops of the mixture of 10 % CaCl2 and 1000 U bovine thrombin to 2mL (milliliter) PRP just before its use in extraction socket.

Surgical procedure The surgical extraction procedure was the same in all patients and carried out by the same operator. After achieving Local anesthesia using 2% lignocaine hydrochloride with 1:100,000 epinephrine, standard Terrence Ward's incision was placed to raise a full thickness mucoperiosteal flap. Distobuccal bone was carefully exposed and bone surrounding the buccal aspect of impacted tooth was performed using surgical bur under copious irrigation with 0.9% saline. The tooth was elevated using Coupland elevator and if required situations tooth was sectioned with surgical bur to facilitate its removal. The socket was checked for any tooth or bony debris. The bony margins smoothened using a file and irrigated with normal saline. Subsequently, PRP gel was placed into the extraction sockets of patients in the group A and wound closure was done using simple interrupted 3.0 black silk sutures. In group B the wound is closed without application of PRP gel. Patients were advised regular post extraction and prescribed 500 mg of paracetamol postoperatively (1 tablet every 6 h for 2 days).

All patients were also advised to not consume any medications but those advised and not to get medical help somewhere else for postoperative discomfort or pain without prior information to the operator. The patients were reviewed postoperatively on 1-, 3-, 5-, 7-, and 14-day to record pain, mouth opening, Soft tissue and bony healing index. Patients were recalled at the 4th, 10th, and 16th postoperative week for assessment of bone healing.

Statistical analysis:

The data were analyzed using SPSS (Statistical Package for the Social Sciences) version 21. Descriptive statistics such as mean, SD (standard deviation ) and percentage were used. Normality of data was tested by using Kolmogorov and Smirnov method. Unpaired t-test was used to compare between groups with normally data and Mann-Whitney test for non-normally data. For categorical variables, Chi-square test was employed. A p-value less than 0.05 were considered as significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients age between 18 and 50 years.
* Patients who required mandibular 3rd molar extractions
* Patients had to have clinical and radiographic diagnosis of a single impacted mandibular third molar
* Radiographic diagnosis of Class II position B impaction (Pell and Gregory classification).
* Patients agree to return for recall visits
* Patients who were not experienced pain, inflammation, and infection at the operating site 7 days before the surgery.

Exclusion Criteria:

Exclusion criterion

* Patients if pregnant, lactating, or smokers or if they had systemic disease or any other medications that could interfere with healing process.
* Any antibiotic or any anti-inflammatory drug usage within a week period.
* Patients with any periapical infection or lesion associated with the third molars
* Patients with unacceptable oral hygiene

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Assessment of pain | 1 week
  Postoperative pain was assessed using a 10-point visual analog scale with a score of 0 equals "no pain" and 10 equals "very severe pain"
Assessment of facial swelling | 1 week
  Facial swelling was assessed by modification of Schultze-Mosgau et al. method, and this involved measuring the length from the tragus to the oral commissure and tragus to the pogonion. The arithmetic sum of the two measurements was considered as facial swelling at the time point.
Assessment of trismus | 1 week
  The maximum distance between the maxillary central incisors and the mandibular central incisors was taken as mouth opening. The difference between postoperative and preoperative mouth opening value was considered as trismus.
Assessment of soft tissue healing | 1 week
  Assessment of soft tissue healing was based on the criteria given by Landry et al. and Gonshor.
Assessment of bone healing | 1 week
  Third molar sockets were assessed radiographically for bone healing by modification of the Kelley's method as described by Olufemi et al.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gawai KT, Sobhana CR. Clinical evaluation of use of platelet rich plasma in bone healing. J Maxillofac Oral Surg. 2015 Mar;14(1):67-80. doi: 10.1007/s12663-013-0605-5. Epub 2014 Jan 9. PMID 25729230
- [Derived] Bailey E, Kashbour W, Shah N, Worthington HV, Renton TF, Coulthard P. Surgical techniques for the removal of mandibular wisdom teeth. Cochrane Database Syst Rev. 2020 Jul 26;7(7):CD004345. doi: 10.1002/14651858.CD004345.pub3. PMID 32712962